CLINICAL TRIAL: NCT01465334
Title: A Phase II Study of Ofatumumab-High Dose Methylprednisolone Followed by Ofatumumab-Alemtuzumab in 17p Deletion CLL
Brief Title: Ofatumumab With High Dose Methylprednisone Followed by Ofatumumab and Alemtuzumab in 17p CLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to change in practice.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Jennifer R. Brown, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-304; NCCN Protocol Number: NCCN-001 (Other Grant/Funding Number: NCCN); GSK Protocol Number: OFT115580 (Other: GSK)
Record Dates: First submitted 2011-10-18; First posted 2011-11-04 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: CLL; SLL
Keywords: 17p Deletion CLL
MeSH Terms: interventions — ofatumumab; Methylprednisolone; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Naive (Experimental): Participants were assigned to 1 of 2 groups based on prior treatment status. Both groups received the same therapy as follows (cycle duration=28 days):
  Induction Part A: Ofatumumab + HDMP 2-4 cycles
  Ofatumumab: cycle 1 - 300 mg intravenously (IV) Day 1 then 1000 mg IV Days 8, 15, 22; cycles 2-4 - 1000 mg IV Days 1, 8, 15, 22
  High-Dose Methylprednisolone (HDMP): 1000 mg/m2 IV Days 1-3
  Participants with nodal complete response at cycle 2 re-staging then discontinued Part A therapy.
  Induction Part B: Ofatumumab + Alemtuzumab 1-6 cycles
  Ofatumumab: 1000 mg IV Day 1
  Alemtuzumab: 30 mg subcutaneously Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24 and 26
  Participants with at least stable disease could continue continue to Part C or, if eligible, proceed to allogeneic stem cell transplant (SCT) off study.
  Maintenance Part C: Ofatumumab + Alemtuzumab up to 26 cycles
  Ofatumumab: 1000 mg IV Day 1 every other cycle
  Alemtuzumab: 30 mg subcutaneously Days 14, 28
  Interventions: Drug: Ofatumumab; Drug: High-Dose Methylprednisolone; Drug: Alemtuzumab
- Relapsed/Refractory (Experimental): Participants were assigned to 1 of 2 groups based on prior treatment status. Both groups received the same therapy as follows (cycle duration=28 days):
  Induction Part A: Ofatumumab + HDMP 2-4 cycles
  Ofatumumab: cycle 1 - 300 mg intravenously (IV) Day 1 then 1000 mg IV Days 8, 15, 22; cycles 2-4 - 1000 mg IV Days 1, 8, 15, 22
  High-Dose Methylprednisolone (HDMP): 1000 mg/m2 IV Days 1-3
  Participants with nodal complete response at cycle 2 re-staging then discontinued Part A therapy.
  Induction Part B: Ofatumumab + Alemtuzumab 1-6 cycles
  Ofatumumab: 1000 mg IV Day 1
  Alemtuzumab: 30 mg subcutaneously Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24 and 26
  Participants with at least stable disease could continue continue to Part C or, if eligible, proceed to allogeneic stem cell transplant (SCT) off study.
  Maintenance Part C: Ofatumumab + Alemtuzumab up to 26 cycles
  Ofatumumab: 1000 mg IV Day 1 every other cycle
  Alemtuzumab: 30 mg subcutaneously Days 14, 28
  Interventions: Drug: Ofatumumab; Drug: High-Dose Methylprednisolone; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Ofatumumab
  Other Names: GSK 1841157
Drug: High-Dose Methylprednisolone
  Other Names: HDMP
Drug: Alemtuzumab
  Other Names: Campath-1H

SUMMARY:
The main purpose of this study is to examine how two separate groups of 17p deletion Chronic lymphocytic leukemia (CLL) participants respond to sequential treatment with this particular combination of drugs. The two groups are those participants who have previously received treatment for their CLL and those who have not yet received any treatment. The combination of drugs is Ofatumumab and High-Dose Methylprednisolone (HDMP) first followed by Ofatumumab and Alemtuzumab. All three drugs are FDA approved and have known activity in treating 17p CLL. We hope that by combining these drugs together in this study, they will have more benefit than each one alone and that the subjects' CLL will be significantly impacted.

DETAILED DESCRIPTION:
Participants were assigned to 1 of 2 groups based on prior treatment status. Both groups received the same therapy.

Part A: Ofatumumab + HDMP 2-4 cycles Part B: Ofatumumab + Alemtuzumab 1-6 cycles Part C: Maintenance with Ofatumumab + Alemtuzumab up to 2 years

Between days 15-22 of Cycle 2 of Part A, participants are restaged. Participants who achieve nodal complete response discontinue Part A therapy and undergo minimal residual disease (MRD) assessment to guide the decision whether to go to Part B or Part C. The participants with persistent disease after 2 cycles of Part A therapy receive 2 more cycles of Part A therapy and then undergo another restaging as well as MRD assessment. At restaging, participants with minimal disease are eligible for Part C or allogeneic stem cell transplant (SCT) off protocol. The remaining participants receive Part B therapy. On Part B, restaging occurs at weeks 12 and 18. If MRD negative complete response (CR) status is achieved then therapy is discontinued and the primary endpoint evaluation occurs 2 months later. Otherwise with persistent disease Part B therapy continues up to 24 weeks and the primary endpoint evaluation occurs after Part B therapy is completed. Participants who achieve clinical complete response may receive Part C therapy or be observed while waiting SCT.

ELIGIBILITY:
Inclusion Criteria:

* Documented CLL/SLL
* 17p deletion by FISH in 20% or more nuclei on peripheral blood, bone marrow or lymph node
* Normal organ function

Exclusion Criteria:

* Pregnant or breast feeding
* Current active hepatic or biliary disease
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, tuberculosis and active Hepatitis C
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* Other past or current malignancy. Participants who have been free of malignancy for at least 2 years, or who have a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible.
* Known HIV positive
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to study entry, congestive heart failure, and arrhythmia unless controlled by therapy, with the exception of extra systoles or minor conduction abnormalities.
* Significant concurrent uncontrolled medical conditions including, but not limited to, renal, hepatic, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease which in the opinion of the investigator may represent a risk for the subject.
* Positive serology for Hepatitis B or C
* History of allergic reactions attributed to ofatumumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R Brown, MD PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davids MS, Kim HT, Yu L, De Maeyer G, McDonough M, Vartanov AR, Langey R, Fernandes SM, Hellman JM, Francoeur K, Arnason J, Jacobsen ED, LaCasce AS, Fisher DC, Brown JR. Ofatumumab plus high dose methylprednisolone followed by ofatumumab plus alemtuzumab to achieve maximal cytoreduction prior to allogeneic transplantation for 17p deleted or TP53 mutated chronic lymphocytic leukemia. Leuk Lymphoma. 2019 May;60(5):1312-1315. doi: 10.1080/10428194.2018.1519814. Epub 2018 Oct 15. PMID 30322319

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled between December 2011 and November 2014.
Period: Overall Study
Arm/Group | Treatment Naive | Relapsed/Refractory
Started | 15 | 15
Complete Part A Induction | 12 | 15
Complete Part B Induction | 7 | 15
Eligible for Allogeneic Transplant | 9 | 9
Completed | 13 | 9
Not Completed | 2 | 6
Not completed — Disease Progression | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Richter's transformation | 0 | 3
Not completed — Refractory Disease | 0 | 3

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Naive | Relapsed/Refractory | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Median (Full Range); unit: years] | 64 [45 to 86] | 65 [58 to 80] | 65 [45 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 10
  Male | 8 | 12 | 20
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30
Number of Prior Therapies [Count of Participants; unit: Participants] — At study entry, participants were classified based on number of prior therapies: treatment naive=0; relapsed/refractory>0.
  Participants
    0 | 15 | 0 | 15
    1 | 0 | 6 | 6
    2 | 0 | 4 | 4
    3 | 0 | 2 | 2
    4 | 0 | 3 | 3
Time from Diagnosis to First Therapy [Mean (Full Range); unit: months] | 6.9 [0.9 to 52.6] | 23 [0.1 to 110] | 12.4 [0.1 to 110]
Time from Diagnosis to Start on Trial [Mean (Full Range); unit: months] | 6.8 [0.8 to 52.6] | 59.4 [1.6 to 233] | 27.6 [0.8 to 233]
Whole Exome Sequencing-Mutations [Median (Full Range); unit: mutations] | 22 [7 to 27] | 20 [15 to 45] | 21 [7 to 45]
Whole Exome Sequencing-Copy Number Alterations [Median (Full Range); unit: Events] | 12.5 [4 to 33] | 14 [3 to 45] | 14 [3 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Induction Overall Response Rate (ORR)
Description: Induction ORR is the percentage of participants achieving a minimum of partial response (PR) over induction treatment based on International Workshop on Chronic Lymphocytic Leukemia (IW-CLL) criteria (Hallek, et al 2008). There are numerous diagnostic tests used for response evaluation including potentially CBC and differential count, marrow aspirate and biopsy, ultrasound of the abdomen, CT scans (chest, pelvis, abdomen) and physical examination. PR is a 50% or greater decrease of measured size of lymphadenopathy, hepatomegaly, splenomegaly as well as blood lymphocytes (over baseline), marrow infiltrate or B-lymphoid nodules and a 50% or greater increase from baseline in platelet count (or level >100,000/micro liter), hemoglobin (or level >11 grams/deciliter), neutrophils (or level >1500/microliter).
Time Frame: Disease was evaluated after weeks 8 and 16 of Part A and at 12, 18 and 24 weeks during part B.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
percentage of participants | 73 [49 to 90] | 60 [36 to 81]

2. Secondary Outcome: Number of Participants Achieving Induction Complete Response (CR)
Description: CR over induction treatment was based on International Workshop on Chronic Lymphocytic Leukemia (IW-CLL) criteria (Hallek, et al 2008). There are numerous diagnostic tests used for response evaluation including potentially CBC and differential count, marrow aspirate and biopsy, ultrasound of the abdomen, CT scans (chest, pelvis, abdomen) and physical examination. CR is absence of significant lymphadenopathy (nodes<1.5 centimeters in long axis diameter), hepatomegaly, splenomegaly as well as blood lymphocytes<4000/microliter, normocellular for age marrow with <30% lymphocytes, no B-lymphoid nodules and platelet>100,000/micro liter, hemoglobin>11 grams/deciliter, neutrophils>1500/microliter.
Time Frame: Disease was evaluated after weeks 8 and 16 of Part A and at 12, 18 and 24 weeks during part B.
Measure: Number; unit: participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
participants | 0 | 0

3. Secondary Outcome: Overall Objective Response Rate (ORR)
Description: Overall ORR is the percentage of participants achieving a minimum of partial response (PR) over induction and maintenance treatment based on International Workshop on Chronic Lymphocytic Leukemia (IW-CLL) criteria (Hallek, et al 2008). There are numerous diagnostic tests used for response evaluation including potentially CBC and differential count, marrow aspirate and biopsy, ultrasound of the abdomen, CT scans (chest, pelvis, abdomen) and physical examination. PR is a 50% or greater decrease of measured size of lymphadenopathy, hepatomegaly, splenomegaly as well as blood lymphocytes (over baseline), marrow infiltrate or B-lymphoid nodules and a 50% or greater increase from baseline in platelet count (or level >100,000/micro liter), hemoglobin (or level >11 grams/deciliter), neutrophils (or level >1500/microliter).
Time Frame: Disease was evaluated after weeks 8 and 16 of Part A, at 12, 18 and 24 weeks during part B and every 6 months on Part C.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
percentage of participants | 80 [56 to 94] | 67 [42 to 86]

4. Secondary Outcome: Number of Participants With Overall CR
Description: CR overall (induction and maintenance treatment) was based on International Workshop on Chronic Lymphocytic Leukemia (IW-CLL) criteria (Hallek, et al 2008). There are numerous diagnostic tests used for response evaluation including potentially CBC and differential count, marrow aspirate and biopsy, ultrasound of the abdomen, CT scans (chest, pelvis, abdomen) and physical examination. CR is absence of significant lymphadenopathy (nodes<1.5 centimeters in long axis diameter), hepatomegaly, splenomegaly as well as blood lymphocytes<4000/microliter, normocellular for age marrow with <30% lymphocytes, no B-lymphoid nodules and platelet>100,000/micro liter, hemoglobin>11 grams/deciliter, neutrophils>1500/microliter.
Time Frame: Disease was evaluated after weeks 8 and 16 of Part A, at 12, 18 and 24 weeks during part B and every 6 months on Part C.
Measure: Number; unit: participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
participants | 2 | 0

5. Secondary Outcome: Overall MRD Negative Rate
Description: Overall MRD negative rate is the percentage of participants classified as MRD negative by four color flow cytometry. The assay has a sensitivity of 1 in 10,000 leukocytes.
Time Frame: MRD was assessed after weeks 8 and 16 of Part A, at 12, 18 and 24 weeks during part B and every 6 months on Part C.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
percentage of participants | 80 [56 to 94] | 53 [30 to 76]

6. Secondary Outcome: Transplant Rate
Description: Percentage of participants eligible for allogeneic hematopoietic stem cell transplantation (alloHSCT) that are able and willing to proceed to alloHSCT.
Time Frame: Evaluated up to 36 cycles (approximately 2.75 years) of treatment (Parts A, B and C)
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
percentage of participants | 43 [21 to 67] | 43 [21 to 67]

7. Secondary Outcome: Number of Participants With Treatment-Related Grades 1-3 Hyperglycemia During Part A Induction
Description: Participants ever experiencing a grade 1-3 hyperglycemia event based on CTCAEv4 with treatment attribution of possible, probably or definite as reported on case report forms were counted.
Time Frame: Adverse Events (AEs) were collected weekly during cycle 1 Part A and then every other week for the duration of Part A (up to 16 weeks)
Measure: Number; unit: participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
participants | 5 | 6

8. Secondary Outcome: 3-Year Progression-Free Survival (PFS) Probability
Description: 3-year PFS is the probability of participants remaining alive and progression-free at 3 years from study entry estimated using Kaplan-Meier methods. Disease progression (PD) per International Workshop on Chronic Lymphocytic Leukemia (IW-CLL) criteria (Hallek, et al 2008) is: the appearance of any new lesion (enlarged lymph node minimum >1.5 centimeters); an increase by 50% in greatest determined diameter of any previous site; an increase in the previously noted enlargement of the liver or spleen by 50% or more or the de novo appearance of hepatomegaly, splenomegaly; a 50% increase of blood lymphocytes (over baseline with level at least 5,000/microliter); occurrence of cytopenia secondary to CLL at least 3 months post treatment including a 50% or greater decrease from baseline in platelet count (or level <100,000/microliter) or a hemoglobin decrease of >2 grams/deciliter (or level <10 grams/deciliter); and transformation to a more aggressive histology.
Time Frame: Disease was evaluated on treatment after weeks 8 and 16 of Part A, at 12, 18 and 24 weeks during part B and every 6 months on Part C as well as off-treatment every 3 months up to 5 years.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
percentage probability | 53 [25 to 74] | 25 [7 to 49]

9. Secondary Outcome: 3-year Overall Survival (OS) Probability
Description: 3-year OS is the probability of participants remaining alive at 3 years from study entry estimated using Kaplan-Meier methods.
Time Frame: Median survival follow-up was 45 months (range 31-58 months) in this study cohort.
Measure: Number (95% Confidence Interval); unit: percentage probability
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
percentage probability | 66 [36 to 84] | 53 [26 to 74]

10. Secondary Outcome: Number of Participants Completing Part A Treatment
Description: Participants counted as completing Part A with either 2 or 4 cycles of treatment per protocol.
Time Frame: Evaluated up to 4 cycles/16 weeks.
Measure: Number; unit: participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
participants | 12 | 15

11. Secondary Outcome: Number of Participants Completing Only 2 Cycles of Part A Treatment
Description: Participants counted if only completed 2 cycles of Part A treatment per protocol.
Time Frame: Evaluated after 2 cycles/8 weeks of Part A therapy.
Measure: Number; unit: participants
Arm/Group | Treatment Naive | Relapsed/Refractory
Number analyzed (Participants) | 15 | 15
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected weekly during cycle 1 Part A and then every other week for the duration of Part A (up to 16 weeks); every cycle for the duration of Part B (up to 24 weeks); and every 56 days for the duration of Part C (up to 104 weeks). AEs in summary were collected up to 144 weeks of treatment plus 30 days.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher. All remaining events regardless of treatment attribution were classified as Other AEs. Grades 1-2 AEs were not required reporting per protocol; all AEs collected were included in the calculation. No further data is available to specify classification of system organ class "Other" per CTCAEv4 criteria beyond the general term.
Groups:
- Treatment Naive; Relapsed/Refractory: Participants were assigned to 1 of 2 groups based on prior treatment status. Both groups received the same therapy.
  (cycle duration=28 days)
  Part A: Ofatumumab + HDMP 2-4 cycles Ofatumumab: 1000 mg IV Days 1, 8, 15, 22 High-Dose Methylprednisolone (HDMP): 1000 mg/m2 IV Days 1-3
  Participants who have not experienced a clinical complete response with no residual detectable disease after Part A will continue on to Part B.
  Part B: Ofatumumab + Alemtuzumab 1-6 cycles Ofatumumab: 1000 mg IV Day 1 Alemtuzumab: 30 mg subcutaneously Days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24 and 26
  Participants who have experienced at least stable disease in Parts A and B can continue on to Part C. Participants who are eligible may instead proceed to stem cell transplantation after Parts A and B.
  Part C: Maintenance with Ofatumumab + Alemtuzumab up to 2 years Ofatumumab: 1000 mg IV every other cycle Alemtuzumab: 30 mg subcutaneously Days 14, 28
Arm/Group | Treatment Naive | Relapsed/Refractory
All-Cause Mortality (participants affected / at risk) | 7/15 | 6/15
Serious Adverse Events (participants affected / at risk) | 11/15 | 9/15
Other Adverse Events (participants affected / at risk) | 15/15 | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Naive (N=15) | Relapsed/Refractory (N=15)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Growth hormone abnormal (Investigations) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Infusion related reaction (General disorders) | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 2
Lymphocyte count increased (Investigations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 6 | 7
Platelet count decreased (Investigations) | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
White blood cell decreased (Investigations) | 4 | 5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Naive (N=15) | Relapsed/Refractory (N=15)
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 3
Alkaline phosphatase increased (Investigations) | 4 | 2
Allergic reaction (Immune system disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 9 | 9
Anorexia (Metabolism and nutrition disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 4 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 9 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 2
Blood bilirubin increased (Investigations) | 2 | 2
Blurred vision (Eye disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Bruising (Injury, poisoning and procedural complications) | 1 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Cardiac disorders - Other (Cardiac disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chills (General disorders) | 4 | 1
Colonic ulcer (Gastrointestinal disorders) | 1 | 1
Confusion (Psychiatric disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Creatinine increased (Investigations) | 2 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Dizziness (Nervous system disorders) | 1 | 0
Dry eye (Eye disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 1 | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 | 0
Edema face (General disorders) | 2 | 0
Edema limbs (General disorders) | 4 | 3
Edema trunk (General disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 0
Eye disorders - Other (Eye disorders) | 2 | 0
Fatigue (General disorders) | 10 | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Fever (General disorders) | 10 | 7
Flashing lights (Eye disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 | 2
General disorders and administration site conditions - Other (General disorders) | 1 | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 4 | 3
Hematoma (Vascular disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6 | 6
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 7 | 4
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2
Infections and infestations - Other (Infections and infestations) | 2 | 0
Infusion related reaction (General disorders) | 3 | 1
Injection site reaction (General disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 4
Investigations - Other (Investigations) | 1 | 0
Irritability (General disorders) | 1 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngitis (Infections and infestations) | 0 | 1
Lipohypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0
Localized edema (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Myelitis (Nervous system disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 0 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nervous system disorders - Other (Nervous system disorders) | 3 | 3
Neutrophil count decreased (Investigations) | 7 | 8
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Papulopustular rash (Infections and infestations) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 2 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 4 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Restlessness (Psychiatric disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 | 3
Skin infection (Infections and infestations) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Superficial thrombophlebitis (Vascular disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 2
Urinary frequency (Renal and urinary disorders) | 4 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Vascular disorders - Other (Vascular disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 3
Weight gain (Investigations) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
White blood cell decreased (Investigations) | 5 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No